CLINICAL TRIAL: NCT01433107
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group Study of the Efficacy and Safety of Terbinafine Film Forming Solution, 1% (as Hydrochloride), in Patients With Tinea Pedis
Brief Title: Efficacy and Safety of Terbinafine Film Forming Solution in Patients With Tinea Pedis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 727-D-301
Record Dates: First submitted 2011-09-08; First posted 2011-09-13 (Estimated); Results first posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Tinea Pedis
Keywords: Tinea pedis; Terbinafine film forming solution
MeSH Terms: conditions — Tinea Pedis | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Terbinafine (Experimental): Drug
  Interventions: Drug: Terbinafine
- Placebo (Placebo Comparator): Drug
  Interventions: Drug: Terbinafine Placebo

INTERVENTIONS:
Drug: Terbinafine — 1% single application
  Arms: Terbinafine
Drug: Terbinafine Placebo — single application
  Arms: Placebo

SUMMARY:
This study will compare the efficacy and safety of a single dose of terbinafine film forming solution 1% with a single dose of placebo film forming solution in the treatment of tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age with interdigital tinea pedis infection, with clinical diagnosis meeting required baseline total sign & symptom score and positive microscopy

Exclusion Criteria:

* Allergy to the allylamine class of antimycotics or excipients in the formulation.
* Chronic, hyperkeratotic plantar (moccasin) tinea pedis
* Other fungal disease or intertrigo
* Other abnormal findings on the affected foot
* Systemic antifungal or antimicrobial treatment within the last 3 months
* Topical treatment for skin lesions on feet within the last 3 months
* Diabetes mellitus and peripheral artery occlusive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking University First Hospital, Beijing
  - Beijing University Hospital N°3, Beijing
  - The Second Affiliated Hospital of Sun Yat-sen University Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Chinese Academy of Medical Sciences, Jiangsu
  - Huashan Hospital, Fudan University, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start 27 Aug 2011 end 14 Feb 2012
Pre-assignment Details: Each particiapant received a single dose of Terbinafine Film Forming Solution 1% or matching placebo
Period: Overall Study
Arm/Group | Terbinafine | Placebo
Started | 145 | 145
Completed | 118 | 128
Not Completed | 27 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terbinafine | Placebo | Total
Number analyzed (Participants) | 145 | 145 | 290
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.27 (12.805) | 34.05 (11.936) | 34.66 (12.372)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 46 | 96
  Male | 95 | 99 | 194

OUTCOME MEASURES:

1. Primary Outcome: Effective Treatment Outcome (Direct Microscopy and Culture Negative and Total Signs and Symptom Score Less or Equal to 2)
Description: Each clinical sign or symptom will be assessed separately. The investigator will evaluate the severity of each sign or symptom over the entire target foot. Clinical signs and symptoms including desquamation (scaling), erythema, incrustation (crusting), pustules, vesiculation and pruritus will be evaluated by the investigator or designee and recorded at every visit using the following scale:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe In order to calculate the total symptoms score the rating for all symptoms are added up.
  Possible range 0 to 18
Time Frame: week 6
Population: Number of success. The discrepancy between number of participants analyzed and participants completed is explained by delayed exclusions (people having negative mycology results received after completion of the study).
Measure: Number; unit: participants
Arm/Group | Terbinafine | Placebo
Number analyzed (Participants) | 115 | 122
participants | 73 | 10

2. Secondary Outcome: Total Clinical Signs and Symptoms (S/S) Scores
Description: Each clinical sign or symptom will be assessed separately. The investigator will evaluate the severity of each sign or symptom over the entire target foot. Clinical signs and symptoms including desquamation (scaling), erythema, incrustation (crusting), pustules, vesiculation and pruritus will be evaluated by the investigator or designee and recorded at every visit using the following scale:
  0 = absent
  1. = mild
  2. = moderate
  3. = severe In order to calculate the total symptom score, the scores for each individual symptom are added up.
  Possible range : 0 to 18
Time Frame: week 6
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Terbinafine | Placebo
Number analyzed (Participants) | 113 | 121
units on a scale | 1.6 [1.3 to 2.0] | 4.7 [4.1 to 5.2]

3. Secondary Outcome: Number of Subjects With Adverse Event
Description: Number of Subjects with adverse event
Time Frame: 6 weeks
Population: Number of subject with any adverse events mild or moderate having signed the informed consent. One subject had an adverse event but did not receive any study drug and was not included in the number of subjects started.
Measure: Number; unit: participants
Arm/Group | Terbinafine | Placebo
Number analyzed (Participants) | 146 | 144
participants | 9 | 11

ADVERSE EVENTS:
Description: One subject had an adverse event but did not receive any study drug and was not included in the number of subjects started.
Arm/Group | Terbinafine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/146 | 0/144
Other Adverse Events (participants affected / at risk) | 0/146 | 7/144
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Terbinafine (N=146) | Placebo (N=144)
General Disorders (General disorders) | 0 (0) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator